CLINICAL TRIAL: NCT04187690
Title: Efficacy and Safety of Jin-shui Huan-xian Granule in the Treatment of IPF
Brief Title: Jin-shui Huan-xian Granule in the Treatment of IPF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TCM for IPF
Record Dates: First submitted 2019-12-03; First posted 2019-12-05 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Idiopathic Pulmonary Fibrosis; traditional Chinese medicine; randomized controlled trial
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Jin-shui Huan-xian granule (Experimental): Participants in this arm will be given Jin-shui Huan-xian granule.
  Interventions: Drug: Jin-shui Huan-xian granule
- Jin-shui Huan-xian granule placebo (Placebo Comparator): Participants in this arm will be given Jin-shui Huan-xian granule placebo.
  Interventions: Drug: Jin-shui Huan-xian granule placebo

INTERVENTIONS:
Drug: Jin-shui Huan-xian granule — Jin-shui Huan-xian granule will be administered 5days on and 2 days off for 52 weeks.
  Arms: Jin-shui Huan-xian granule
Drug: Jin-shui Huan-xian granule placebo — Jin-shui Huan-xian granule placebo will also be administered 5days on and 2 days off for 52 weeks. The placebo consists 5% of the same components as Jin-shui Huan-xian granule besides dextrin and bitter. The There is no obvious difference in appearance, weight and odor between Jin-shui Huan-xian granule and placebo.
  Arms: Jin-shui Huan-xian granule placebo

SUMMARY:
This study is to evaluate the efficacy and safety of Jin-shui Huan-xian granule for idiopathic pulmonary fibrosis (IPF), establish the treatment scheme, and obtain the high quality clinical evidences.

DETAILED DESCRIPTION:
Idiopathic pulmonary fibrosis (IPF) is a chronic, progressive and ultimately fatal interstitial lung disease. With worsened dyspnea and an increasing loss of pulmonary function, IPF patients will have very poor quality of life. It has also brought an increasing social-economic burden. Researches show that pirfenidone and nintedanib could be effective to IPF, which were also recommended by the guideline. However, the application has been limited by side effects and high prices. It is urgent to develop other effective treatments and strategies to manage IPF. The investigators' previous studies shown that Jin-shui Huan-xian granule could be effective to IPF.

This is a multicerter, randomized, double-blind, placebo-controlled trial to assess the efficacy of Jin-shui Huan-xian granule in reducinig the acute exacerbations, improving exercise capacity, and delaying the disease progression for IPF. After a 2-week wash-out period, 312 patients will be randomly assigned into treatment or control group for 52-week treatment. The primary outcomes are frequencies of acute exacerbation, 6-minute walking test, and percentage of patients with progression-free survival. The secondary outcomes include pulmonary function, all-cause mortality, clinical symptoms, dyspnea score, and quality of life. Safety will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* A confirmed diagnosis stable IPF.
* Age ranges from 40 years to 85 years.
* TCM Syndrome differentiation meets criteria of pattern of Lung Qi deficiency, yin deficiency and inter heat, and lung-kidney qi deficiency.
* Without participanting in any other trial.
* With signed informed consent.

Exclusion Criteria:

* Pregnant, nursing or may become pregnant women.
* Patients with unconscious, dementia or mental disorders.
* Patients with severe cardiac dysfunction.
* Patients with severe liver and kidney diseases.
* Patients with asthma, bronchiectasis, active pulmonary tuberculosis, pulmonary embolism, chronic obstructive pulmonary disease, chronic respiratory failure or other severe respiratory diseases.
* Patients with tumor after resection, radiotherapy or chemotherapy in the past 5 years.
* Patients with severe neuromuscular disorders, severe arthritis or severe peripheral vascular diseases.
* Patients with long-term bedridden.
* Patients who are allergic to any of the treatment drugs.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Frequencies of acute exacerbations (AEs) | up to 52 weeks.
  It will be assessed by frequencies of AEIPF-related hospitalizations.
Six-minute walking distance(6MWD) | Change from baseline 6MWD at week 13, 26, 39 and 52
  6MWD will be applied to evaluate the exercise capacity. The higher values indicate the better exercise capacity.
Proportion of progressive-free survival | up to week 13, 26, 39 and 52.
  Endpoints of Progressive-free survival include FVC decreased by 10% compared with baseline, or DLCO% decreased by 15%, or death or lung transplantation.

SECONDARY OUTCOMES:
Pulmonary function | Change from baseline FVC and DLco% at week 26 and 52.
  Forced vital capacity (FVC) and diffusing capacity percentage of the predicted value (DLco%) will be applied to assess pulmonary function.
All-cause mortality | up to 52 weeks.
  The all-cause mortality will be calculated in each group at the end of the trial.
Clinical symptoms and Signs | Change from baseline clinical symptoms assessment questionnaire scores at week 13, 26, 39 and 52.
  Assessment will be performed by clinical symptom assessment questionnaire. The clinical symptoms to be evaluated in this study include cough, expectoration, chest tightness, shortness of breath, wheezing and cyanosis. A score of 0-3 will be given to every symptom or sign with a higher score indicating a worse conditoin.
Dyspnea | Change from baseline mMRC scores at week 13, 26, 39 and 52.
  Dyspnea will be assessed by modified Medical Research Council (mMRC) scores set up by American Thoracic Society. A score of 0-4 will be given according to the degree of immediate dyspnea. A higher score indicates a worse dyspnea.
COPD assessment test (CAT) | Change from baseline CAT scores at week 13, 26, 39 and 52.
  CAT will be used to evaluate quality of life. A total score of 0-40 will be given with a higher score indicating a worse condition.
36-item short-form health survey (SF-36) total scores | Change from baseline SF-36 scores at week 13, 26, 39 and 52.
  SF-36 total scores will be used to evaluate quality of life with a total score of 0-100. The higher scores will indicate the better outcomes.
St. George's respiratory questionnaire (SGRQ) total scores | Change from baseline SGRQ scores at week 13, 26, 39 and 52.
  SGRQ total scores will be used to evaluate quality of life with a total score of 0-100. The higher scores will indicate the worse outcomes.
A Tool to Assess Quality of life in IPF(ATAQ-IPF) | Change from baseline ATAQ scores at week 13, 26, 39 and 52.
  ATAQ-IPF will be used to evaluate quality of life. There are 13 domains with 74 items with a score of 1-5 for each item. A higher score will indicate a worse health.

CONTACTS AND LOCATIONS:
Overall Officials: Jian-sheng Li, Professor, Study Chair — The First Affiliated Hospital of Henan University of Traditional Chinese Medicine
Locations (1):
- the First Affiliated Hospital of Henan University of Chinese Medicine, Zhengzhou, China

REFERENCES:
- [Derived] Yang SG, Yu XQ, Li JS, Xie Y, Zhang W, Ban C, Feng J, Wu L, Lu X, Zhao L, Meng Y, Zhou M, He Y, Luo W. Efficacy and safety of Jin-shui Huan-xian granule for idiopathic pulmonary fibrosis: study protocol for a multicenter, randomized, double-blind, placebo-controlled trial. Trials. 2022 Sep 2;23(1):725. doi: 10.1186/s13063-022-06684-0. PMID 36056382